CLINICAL TRIAL: NCT04851392
Title: Do Adolescents and Adults Differ in Their Acute Subjective, Behavioural and Neural Responses to Cannabis, With and Without Cannabidiol?
Brief Title: Do Adolescents and Adults Differ in Their Acute Response to Cannabis?
Acronym: CannTeenA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); Invicro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 5929/005
Record Dates: First submitted 2021-04-05; First posted 2021-04-20 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cannabis; Cannabis Intoxication; Cannabis Use; Cannabis Dependence; Marijuana; THC; CBD; Adolescent Development
Keywords: Cannabis; Marijuana; THC; CBD; Adolescence; fMRI; Cognition; Subjective effects; Psychotomimetic effects
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol; Cannabidiol

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, crossover experiment with drug condition block randomised and stratified by age-group and gender, such that drug order is counterbalanced.
  There are two groups: adolescents (16-17 years old) and adults (26-29 years old). These groups are matched on current cannabis use frequency.
  There are three drug conditions: (1) cannabis with delta-9-tetrahydrocannabinol (THC) and without cannabidiol (CBD), (2) cannabis with THC but without CBD, and (3) placebo cannabis without THC and without CBD.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- THC condition (Experimental): THC condition: Cannabis with delta-9-tetrahydrocannabinol (THC) and no cannabidiol (CBD). 0.107mg/kg of THC. A 75kg person receives 8mg of THC.
  Route of administration: vaporised and inhaled.
  Frequency: once.
  Duration: inhaled in < 18 minutes.
  Interventions: Drug: Cannabis with delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD)
- THC+CBD condition (Experimental): THC+CBD condition: Cannabis with THC and CBD (i.e. THC+CBD condition). 0.107mg/kg of THC and 0.320mg/kg of CBD. A 75kg person receives 8mg of THC and 24mg of CBD.
  Route of administration: vaporised and inhaled.
  Frequency: once.
  Duration: inhaled in < 18 minutes.
  Interventions: Drug: Cannabis with THC without CBD
- PLA condition (Placebo Comparator): PLA condition: Placebo cannabis with no THC or CBD.
  Route of administration: vaporised and inhaled.
  Frequency: once.
  Duration: inhaled in < 18 minutes.
  Interventions: Drug: Placebo cannabis

INTERVENTIONS:
Drug: Cannabis with delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) — Cannabis with delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) - inhaled and vaporised cannabis flower
  Arms: THC condition
Drug: Cannabis with THC without CBD — Cannabis with THC without CBD - inhaled and vaporised cannabis flower
  Arms: THC+CBD condition
Drug: Placebo cannabis — Placebo cannabis, without THC and without CBD - inhaled and vaporised
  Arms: PLA condition

SUMMARY:
The acute effects of cannabis may differ between adolescents and adults. Furthermore, these effects may be tempered by the presence of cannabidiol. This double-blind, placebo-controlled, crossover experiment investigates the acute effects of cannabis (with and without cannabidiol) on subjective effects, behavioural responses and neural functioning in 16-17 year-olds and 26-29 year-olds who regularly use cannabis (0.5-3 days per week).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents: Aged 16-17
* Adults: Aged 26-29 years
* Self-reported cannabis use between 0.5 and 3 days/week, averaged over the last 3 months
* Adults: Body mass index (BMI) between 18.5 and 29.9
* Adolescents: BMI between 2nd percentile and 98th percentile
* Self-reported ability to consume approximately half a typical joint of cannabis by themselves within 20 minutes
* Willing to be cannulated and have four blood samples taken at every acute session
* Right-handed

Exclusion Criteria:

* Females: Pregnant or breast-feeding
* Adults: Before the age of 18, had a period of 3 or more months when cannabis was used once per week or more frequently.
* Severe cannabis use disorder (DSM-5)
* Illicit drug use of any specific drug more than twice per month, averaged over the last 3 months
* Receiving treatment (pharmacological or psychological) for a mental health problem within the last month
* Lifetime psychosis
* Lifetime psychosis of any immediate family member
* Hypertension (systolic > 160 or diastolic > 100)
* Dependent on tobacco or vaping nicotine (> 1 on the Heaviness of Smoking Index)
* Currently taking a psychotropic medication that will likely affect dependent variables or interact with cannabis
* Any physical or mental health condition, any medication, or any treatment, that the study doctor considers to be an exclusion
* MRI contraindications
* Significant asthma or respiratory problems - severity judged clinically
* Self-reported moderate/severe acute unpleasant effects from cannabis which occur often or always
* Positive alcohol breathalyser reading at any acute session (rearrange session)
* Self-reported use of alcohol within 24 hours at any acute session (rearrange session)
* Self-reported use of illicit drugs (including cannabis) within 72 hours at any acute session (rearrange session)
* Positive saliva drug screen at any acute session (rearrange session)

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Psychotomimetic effect | Measured once, 2 hours after the start of drug administration, on each drug condition
  Measured by total Psychotomimetic States Inventory (PSI) score
Verbal episodic memory | Measured once, 2 hours after the start of drug administration, on each drug condition
  Measured by delayed prose recall performance
Strength of subjective drug effect | Measured 20 minutes after the start of drug administration, on each drug condition
  Measured by self-reported 'feel drug effect', rated from 0 (not at all) to 10 (extremely)

SECONDARY OUTCOMES:
Self-reported subjective effects | Measured -30 minutes, 20 minutes, 30 minutes, 2 hours, and 2 hours & 40 minutes after the start of drug administration, on each drug condition
  Feel drug effect, like drug effect, dislike drug effect, alert, want to have cannabis, happy, relaxed, anxious, paranoid, mentally impaired, stoned, dry mouth, unmotivated, intensified sensory perception, want to listen to music, want food, want to see friends, rated from 0 (not at all) to 10 (extremely)
Functional magnetic resonance imaging (fMRI) measured neural correlates | Measured between 40 minutes and 1 hour & 20 minutes after the start of drug administration, on each drug condition
  Reward anticipation and reward feedback, response inhibition, spatial working memory, and resting-state
Magnetic resonance spectroscopy | Measured 1 hour & 30 minutes after the start of drug administration, on each drug condition
  Measuring glutamate levels in the dorsal striatum
Positive and negative syndrome scale | Measured 2 hours & 40 minutes after the start of drug administration, on each drug condition
  Kay et al. (1987). Higher scores reflect stronger positive and negative symptoms.
Effort-related decision-making (i.e. amotivation) | Measured 2 hours & 20 minutes after the start of drug administration, on each drug condition
  Measured by the physical effort task ('apple-gathering' task) as described in Husain & Roiser (2018)
Pleasure processing | Measured 2 hours & 30 minutes after the start of drug administration, on each drug condition
  Measured by subjective liking in response to chocolate, music and cartoons, rated from 0 (not at all) to 10 (extremely), similar to Lawn et al. (2015)
Visual attentional bias to cannabis and food stimuli | Measured 2 hours & 10 minutes after the start of drug administration, on each drug condition
  Measured by the visual dot-probe task, as described in Morgan et al. (2010)
Heart rate | Measured -30 minutes, 20 minutes, 30 minutes, 2 hours, and 2 hours & 40 minutes after the start of drug administration, on each drug condition
  Measuring heart rate
Blood pressure | Measured -30 minutes, 20 minutes, 30 minutes, 2 hours, and 2 hours & 40 minutes after the start of drug administration, on each drug condition
  Measuring systolic and diastolic blood pressure.
Exogenous and endogenous cannabinoid levels in plasma | Measured -30 minutes, 20 minutes, 30 minutes, and 2 hours & 40 minutes after the start of drug administration, on each drug condition
  Measuring THC and CBD and metabolites; and endocannabinoids
Dissociative states scale | Measured 2 hours & 40 minutes after the start of drug administration, on each drug condition
  Bremner et al. (1998). Higher scores reflect greater dissociation.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall D, Lawn W, Ofori S, Trinci K, Borissova A, Mokrysz C, Petrilli K, Bloomfield MAP, Wall MB, Freeman TP, Curran HV. The acute effects of cannabis, with and without cannabidiol, on attentional bias to cannabis related cues: a randomised, double-blind, placebo-controlled, cross-over study. Psychopharmacology (Berl). 2024 Jun;241(6):1125-1134. doi: 10.1007/s00213-024-06543-7. Epub 2024 Feb 28. PMID 38416223
- [Derived] Lawn W, Trinci K, Mokrysz C, Borissova A, Ofori S, Petrilli K, Bloomfield M, Haniff ZR, Hall D, Fernandez-Vinson N, Wang S, Englund A, Chesney E, Wall MB, Freeman TP, Curran HV. The acute effects of cannabis with and without cannabidiol in adults and adolescents: A randomised, double-blind, placebo-controlled, crossover experiment. Addiction. 2023 Jul;118(7):1282-1294. doi: 10.1111/add.16154. Epub 2023 Feb 26. PMID 36750134
- [Derived] Skumlien M, Freeman TP, Hall D, Mokrysz C, Wall MB, Ofori S, Petrilli K, Trinci K, Borissova A, Fernandez-Vinson N, Langley C, Sahakian BJ, Curran HV, Lawn W. The Effects of Acute Cannabis With and Without Cannabidiol on Neural Reward Anticipation in Adults and Adolescents. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 Feb;8(2):219-229. doi: 10.1016/j.bpsc.2022.10.004. Epub 2022 Oct 28. PMID 36642667
- [Derived] Dhami P, Quilty LC, Schwartzmann B, Uher R, Allen TA, Kloiber S, Lam RW, MacQueen G, Frey BN, Milev R, Muller DJ, Strother SC, Blier P, Soares CN, Parikh SV, Turecki G, Foster JA, Rotzinger S, Kennedy SH, Farzan F. Response Inhibition and Predicting Response to Pharmacological and Cognitive Behavioral Therapy Treatments for Major Depressive Disorder: A Canadian Biomarker Integration Network for Depression Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 Feb;8(2):162-170. doi: 10.1016/j.bpsc.2021.12.012. Epub 2022 Jan 13. PMID 35032682